CLINICAL TRIAL: NCT02383875
Title: An Interventional Study to Reduce Social Disparities in Diet Quality in the Northern Districts of Marseille (Opticourses)
Brief Title: An Interventional Study to Reduce Social Disparities in Diet Quality in the Northern Districts of Marseille
Acronym: Opticourses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Principal Investigator, Nicole Darmon, PhD, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Opticourses
Record Dates: First submitted 2015-02-25; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Nutritional Quality of Food Purchases
Keywords: nutrition economics; food expenditure; nutritional quality; low income

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Opticourses education intervention (Experimental): People living in the northern districts of Marseille with in very deprived social situation: very low incomes, heavy financial dependence on social benefits, over-representation of people covered by arrangements for controlling poverty and people covered by free social security
  Interventions: Behavioral: Opticourses

INTERVENTIONS:
Behavioral: Opticourses — An intervention session consisted of five two-hour educative workshops which aimed to help people to improve the nutritional quality of food purchases under budgetary constraints.

SUMMARY:
The Opticourses project aims to improve the nutritional quality/price (NQP) ratio of the food purchases of people claiming to be facing financial problems. Following one of the main principles of the French National Nutrition and Health Program (PNNS), the project starts from the principle that to modify food consumption favourably and durably, one must act on both the demand and the supply (see figure). The "demand" part of the project is based on participatory workshops, and the "supply" part relies on intervention of social marketing in shops.

DETAILED DESCRIPTION:
The demand part of the project is based on intervention sessions consisting in five two-hour workshops with about ten participants. The workshops were based on the people's actual purchases and notably on their till receipts. During the five sessions, the receipts were used as intervention tools: participants and research staff discussed the receipts brought in by them all, and exchanged ideas and experiences around food purchasing behaviors.

* First workshop: Opticourses intervention presentation, discussion about grocery shopping strategies, explanation of protocol for receipt collection and annotation, two quiz on nutritional knowledge, food shopping exercise on a catalog;
* Second workshop: discussion about the receipt collection and help to participants encountering difficulties, food groups teaching;
* Third workshop: till receipts delivery by each participant, food with a high nutritional quality for their price teaching;
* Fourth workshop: individual return on the nutritional quality of food purchase on the basis of till receipts analysis, individual objectives to improve the nutritional quality of food purchase at no additional cost, discussion about discount food representations, two quiz on nutritional knowledge, food shopping exercise on a catalog;
* Fifth workshop: assessment of the Opticourses intervention with the participants, discussion about their behavioral modification regarding grocery shopping.

The supply part of the project aims at influencing the supply by means of social marketing. The research team intervenes in two "discount" shops (DIA retailer) in the northern districts in order to influence the food supply. In collaboration with the agency Link Up, a specialist in social marketing, a campaign to promote foods with a good NQP ratio has been launched (from January until June 2014). This public health campaign has the aim of making good NQP foods visible, available and attractive. For 6 months, all the foods with a good NQP ratio in the shop (identified by the research team) are put at the front of the shelves. Consumers can spot them thanks to a logo, "EAT TOP", accompanied by the claim "Nutritious and inexpensive; that's TOP". Good NQP foods are presented with the support of flyers and recipes, simple and accessible to everyone. Also, placing at the head of the gondola and in-store exhibitions are planned around star foods of the month. During the first two months, fish and canned foods will be given the most prominence. Consumers will find in the flyers made available: nutritional information, tips and tricks for cooking them, simple cheap recipes (less than 1€ per person) combining these good NQP foods (sardine rillettes, tuna pâté, etc.) and a TOP selection of good NQP foods available in the store.

ELIGIBILITY:
Inclusion Criteria:

* living in the northern districts of Marseille
* willingness to be involved in an intervention session aimed at improving the nutritional quality of food purchases under budgetary constraints

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic of nutritional quality of food purchases | One-month - Between the first and the third workshop
  Opticourses participants collected food purchase receipts for their household over a one-month period which constituted a detailed record of the quantities of food entering their household. They were asked to save all till receipts for foods consumed at home. To facilitate data collection, participants were given a notebook of food purchases in which they could find step-by-step instructions, example receipts, and, on the last page, an envelope in which to collect the receipts. In case of incomplete or ambiguous printed information regarding the name of the shop, the name of a food, the quantities purchased or the price paid for a food, participants were instructed to write it on the receipt. Expenditure without receipts (gifts or other sources) was to be recorded in the notebook. The participants were also requested to ask other household members to keep their till receipts.

SECONDARY OUTCOMES:
Nutritional knowledge assessment: food groups | At the first workshop and 6 weeks later at the fourth
  At the first workshop, Opticourses participants had to answer a quiz about food groups in order to assess their knowledge prior to the Opticourses intervention. At the fourth workshop, they answered the same quiz which permitted us to measure the intervention effect.
Nutritional knowledge assessment: food with a high nutritional quality for their price | At the first workshop and 6 weeks later at the fourth
  At the first workshop, Opticourses participants had to answer a quiz about their knowledge of what is a food with a high nutritional quality for its price prior to the Opticourses intervention. At the fourth workshop, they answered the same quiz which permitted us to measure the intervention effect.
Experimental economics: food purchases on catalog | At the first workshop and 6 weeks later at the fourth
  At the first workshop, Opticourses participants were asked to shop for food for two days and for all the members of their household on the basis of a food catalog. This catalog included food items with different price options. At the fourth workshop, they did it once again which permitted it to evaluate the intervention effect on their purchase intention regarding nutritional quality and price.

REFERENCES:
- [Derived] Tharrey M, Dubois C, Maillot M, Vieux F, Mejean C, Perignon M, Darmon N. Development of the Healthy Purchase Index (HPI): a scoring system to assess the nutritional quality of household food purchases. Public Health Nutr. 2019 Apr;22(5):765-775. doi: 10.1017/S1368980018003154. Epub 2018 Nov 26. PMID 30472975
- [Derived] Perignon M, Dubois C, Gazan R, Maillot M, Muller L, Ruffieux B, Gaigi H, Darmon N. Co-construction and Evaluation of a Prevention Program for Improving the Nutritional Quality of Food Purchases at No Additional Cost in a Socioeconomically Disadvantaged Population. Curr Dev Nutr. 2017 Sep 13;1(10):e001107. doi: 10.3945/cdn.117.001107. eCollection 2017 Oct. PMID 29955680
- [Derived] Marty L, Dubois C, Gaubard MS, Maidon A, Lesturgeon A, Gaigi H, Darmon N. Higher nutritional quality at no additional cost among low-income households: insights from food purchases of "positive deviants". Am J Clin Nutr. 2015 Jul;102(1):190-8. doi: 10.3945/ajcn.114.104380. Epub 2015 May 27. PMID 26016868
- See also: Opticourses project website — http://www.opticourses.fr/